CLINICAL TRIAL: NCT06599073
Title: A Feasibility Study to Evaluate a New Doppler Method (RescueDoppler) for Monitoring Blood Flow in the Carotid Artery in Subjects Suffering From Sudden Cardiac Arrest
Brief Title: RescueDoppler- a Disruptive Ultrasound Solution for Improved Outcome After Cardiac Arrest.
Acronym: RescueDoppler
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Nordlandssykehuset HF (Other); Ullevaal University Hospital (Other); Rikshospitalet University Hospital (Other); University Hospital, Akershus (Other); Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 582681; 332205 (Other Grant/Funding Number: The Research Council of Norway)
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Cardiac Arrest (CA); Cardiopulmonary Resuscitation; Doppler Ultrasound
Keywords: Continuous ultrasound during cardiac arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RescueDoppler patch with probe is attached to patients with cardiac arrest (Experimental): The RescueDoppler probe and patch are placed on the left side of the patient's neck in both pre-hospital and in-hospital settings. The RescueDoppler system is blinded to the medical personnel during the cardiac arrest and is not used for real-time monitoring. After the cardiac arrest, the velocity curves are processed by the research team and synchronized with the ECG for analysis.
  Interventions: Device: RescueDoppler; Device: Rescue

INTERVENTIONS:
Device: RescueDoppler — Continuous hands-free Doppler ultrasound of the carotid artery during cardiac arrest
  Other Names: Carotid Doppler
Device: Rescue — RescueDoppler patch with probe is attached on the left side of the neck during the cardiac arrest. Operative health personell are blinded for the velocity curves that are post-processed by the research team after the cardiac arrest and synchronised with ECG.

SUMMARY:
RescueDoppler is an innovative, hands-free Doppler system designed for continuous monitoring of blood flow in the carotid artery, distinguishing between the presence and absence of a pulse. It is non-invasive, user-independent, and does not require specialized ultrasound expertise. The primary goal of this study is to assess the feasibility and clinical utility of RescueDoppler for monitoring carotid artery blood flow in patients experiencing sudden cardiac arrest.

The multi-center study will be performed both pre-hospital and in-hospital.

DETAILED DESCRIPTION:
When treating sudden cardiac arrest (SCA), manual pulse checks are currently the standard method to detect blood flow, but this approach has significant limitations. It's neither quick nor consistently reliable (Germanoska et al. 2018, Eberle et al. 1996). Studies show that 45% of healthcare workers struggle to accurately detect a central pulse during cardiac arrest (Moule 2000, Nakagawa et al. 2010). If blood flow has already been restored, continuing chest compressions could cause more harm than good. This highlights the need for an easy-to-use tool to assess blood flow during cardiopulmonary resuscitation (CPR).

Cardiac arrest is responsible for 7-8 million deaths per year and ranks as the third leading cause of death in industrialized countries. Despite advances in resuscitation techniques and post-resuscitation care, the survival rate following cardiac arrest remains low-around 10% or less. Survival rates drop sharply with every minute that passes without advanced cardiac life support (OECD 2017). Successful resuscitation after cardiac arrest requires restoring the heart's normal electrical activity and ensuring adequate blood flow to vital organs. Currently, only the heart's electrical activity (via electrocardiogram [ECG]) is monitored during resuscitation, with no information available on blood flow.

CPR involves chest compressions and artificial ventilation to maintain circulation and oxygenation. In cases of shockable rhythms, a defibrillator delivers an electrical shock to the heart. Automated external defibrillators (AEDs) are capable of diagnosing life-threatening arrhythmias, enabling even untrained bystanders to use them effectively. However, while defibrillators can detect, treat, and confirm the return of normal heart rhythm, they don't provide feedback on whether blood flow has been successfully restored (return of spontaneous circulation [ROSC]). A quicker ROSC is linked to better long-term survival outcomes.

Non-shockable rhythms, such as pulseless electrical activity (PEA) and asystole, are increasingly common. Research shows that up to 60% of patients with suspected PEA and 10-35% of those with suspected asystole still have mechanical heart activity (Deakin 2000, Gaspari et al. 2016). In these cases, using cardiac ultrasound has changed patient management in 78% of cases and has been linked to increased survival. European Resuscitation Council guidelines recommend limiting interruptions during CPR to 10 seconds to check for a pulse (Perkins et al. 2021). However, cardiac ultrasound cannot be performed during chest compressions, which limits its usefulness (Zengin et al. 2018).

Doppler ultrasound measurements of carotid artery blood flow offer a promising alternative for guiding CPR without interrupting resuscitation. The RescueDoppler system, a newly developed ultrasound Doppler tool, continuously monitors blood flow in the carotid artery during CPR.

The RescueDoppler device uses a small ultrasound probe that is quickly attached over the carotid artery using an innovative patch. This probe continuously monitors blood flow to the brain, alerting first responders if chest compressions are ineffective or if the patient has achieved ROSC (when the heart starts beating again).

RescueDoppler probe is placed on the left side of the neck during cardiac arrest to monitor blood flow from the carotid artery during CPR. The medical team won't see the signals during this phase.

The multi-centre study will involve 300 patients experiencing in-hospital or pre-hospital cardiac arrests. Five hospitals in Norway will participate in the in-hospital portion, with recruitment expected to take one year. The pre-hospital study will include two hospitals in Norway, also with a one-year recruitment period. The goal is to gather crucial medical and physiological data on blood circulation during cardiac arrest, beyond initial feasibility.

ELIGIBILITY:
Inclusion Criteria:

Male or female, aged 18 years or older. Subjects experiencing a sudden cardiac arrest, either pre-hospital or in-hospital. Sudden cardiac arrest is defined as the abrupt loss of heart function, breathing, and consciousness.

Exclusion Criteria:

Subjects where resuscitation is not continued after the initial application of RescueDoppler or resuscitation efforts are halted due to a do-not-resuscitate order.

Subjects deemed unable to comply with the study requirements as determined by the Investigator.

Subjects with extensive trauma injuries that prevent proper attachment of the RescueDoppler patch.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with carotid peak blood flow velocity of more than 20 cm/second during cardiopulmonary resuscitation | From enrollment to the end after 12 months
  A carotid peak blood flow velocity of zero indicates the absence of spontaneous circulation during cardiopulmonary resuscitation, while velocities exceeding 20 cm/second suggest the presence of spontaneous circulation.

SECONDARY OUTCOMES:
Number of patients with carotid peak blood flow velocity of more than 50 cm/second during chest compressions | From enrollment to the end after 12 months
  A carotid peak blood flow velocity of zero indicates ineffective chest compressions, while velocities exceeding 50 cm/second suggest that the chest compressions are effective.

CONTACTS AND LOCATIONS:
Locations (8):
- Norway (7):
  - Akershus university hospital, Loerenskog, Akershus
  - Haukeland University Hospital, Surgical Services Clinic, Department of Emergency Medicine, Bergen, Vestland
  - Nordland Hospital, Bodø
  - Oslo University Hospital Ullevål location Lørenskog, Oslo
  - Oslo University Hospital Rikshospitalet, Oslo
  - Oslo University Hospital Ullevaal, Oslo
  - St Olavs University Hospital, Trondheim
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
ECG and carotid blood flow velocity will be shared if required.
Supporting Information: ICF, CSR
Time Frame: Starting 6 months after the publication of results and ending 2 years later.
Access Criteria: A data sharing agreement must be signed and submitted to the steering committee, which includes the Principal Investigator (PI) and Site Investigators (SI) from all participating hospitals in the study.

REFERENCES:
- [Result] Faldaas BO, Nielsen EW, Storm BS, Lappegard KT, Nilsen BA, Kiss G, Skogvoll E, Torp H, Ingul CB. Real-time feedback on chest compression efficacy by hands-free carotid Doppler in a porcine model. Resusc Plus. 2024 Feb 20;18:100583. doi: 10.1016/j.resplu.2024.100583. eCollection 2024 Jun. PMID 38404755
- [Result] Faldaas BO, Nielsen EW, Storm BS, Lappegard KT, How OJ, Nilsen BA, Kiss G, Skogvoll E, Torp H, Ingul C. Hands-free continuous carotid Doppler ultrasound for detection of the pulse during cardiac arrest in a porcine model. Resusc Plus. 2023 Jun 20;15:100412. doi: 10.1016/j.resplu.2023.100412. eCollection 2023 Sep. PMID 37448689
- See also: RescueDoppler website — https://www.rescuedoppler.com